CLINICAL TRIAL: NCT02211339
Title: An Investigation Into the Effectiveness of a Social Communication Skills Training Programme for Adults Following Brain Injury Using a Peer Learning Model
Brief Title: A New Intervention for Social Communication Skills Following Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCL JRO ref: 13/0477; 14/SC/0048 (Other: South Central Hampshire 'A' Research Ethics Committee)
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Brain Injuries
Keywords: Social skills; Social communication; Cognitive communication; Traumatic brain injury; Acquired brain injury; Communication partner training; Peer partner training; Peer mentoring; Rehabilitation
MeSH Terms: conditions — Brain Injuries; Social Skills; Communication; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: An experimental parallel group design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-led intervention group (Experimental): Individuals met twice a week for 8 weeks and participated in a peer-mediated social communication skills group.
  Interventions: Behavioral: Peer facilitator training
- Staff-led social activity group (Active Comparator): Individuals met twice a week for 8 weeks and participated in staff-led social activities.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Peer facilitator training — Peer facilitation of a project-based activity without staff present
  Arms: Peer-led intervention group
Other: Usual care — Staff-led social activity
  Arms: Staff-led social activity group

SUMMARY:
To investigate the effectiveness of a peer-led social skills training intervention compared to social activity (usual care) to improve social communication skills following severe brain injury.

DETAILED DESCRIPTION:
A pilot study first tested the feasibility of the approach and the sensitivity of existing outcome measures to changes in group social interaction. Following amendments to the pilot protocol, twelve new participants with severe ABI were recruited from a residential post-acute rehabilitation centre in April 2015. An experimental parallel group design was used to compare a peer-led group intervention to a staff-led social activity group. Participants were randomised to a peer-led intervention (n=6) or a staff-led social activity group (usual care) (n=6). The groups met twice a week for 8 weeks. A peer with severe ABI was trained separately to facilitate interaction in the peer-led group. The training took place in 16 individual sessions over 4 weeks. Group behaviour was measured twice at baseline, after intervention and at maintenance (4 weeks) using measures meeting reliability, validity and responsiveness criteria tested in the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 70 years
* A diagnosis of severe traumatic brain injury (TBI) or severe acquired brain injury (ABI) with similar cognitive presentation to TBI
* Minimum of six months post injury
* Evidence of a social communication impairment as a result of injury
* Ability to tolerate group activity

Exclusion Criteria:

* Significant aphasia
* Severe depression or psychiatric disorder
* Insufficient English to converse with peers
* Profound cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The Adapted Measure of Participation in Conversation (MPC): Interaction Scale | Baseline to maintenance (week 12)
  This 9 point Likert scale is a measure of verbal and non-verbal participation in conversation. Scores range from 0 (no participation) to 4 (full participation) with half point scoring.
The Adapted Measure of Participation in Conversation (MPC): Transaction Scale | Baseline to maintenance (week 12)
  This 9 point Likert scale is a measure of the ability to share and request information in conversation. Scores range from 0 (no participation) to 4 (full participation) with half point scoring.
The Interactional Network Tool (INT) | Baseline to maintenance (week 12)
  A new measure of group social participation developed for this study. The INT captures group interaction patterns using communication behaviour frequencies and principles of social network analysis. The data is relational and follows a scale-free distribution.

SECONDARY OUTCOMES:
La Trobe Communication Questionnaire (LCQ) (self-report) | Baseline to maintenance (week 12)
  A 30 item self-report questionnaire measuring perceived change in social communication skills. Response options are entered on a four point Likert scale (range: 30-120 with a higher score indicating more impaired skills).
La Trobe Communication Questionnaire (LCQ) (other-report) | Baseline to maintenance (week 12)
  A 30 item questionnaire measuring perceived change in social communication skills, rated by a familiar communication partner. Response options are entered on a four point Likert scale (range: 30-120 with a higher score indicating more impaired skills).

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Beeke, PhD, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: Yes
Available on request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting after publication (2019)
Access Criteria: University College London open access repository
URL: http://discovery.ucl.ac.uk

REFERENCES:
- [Derived] Howell S, Beeke S, Pring T, Varley R. Measuring outcomes of a peer-led social communication skills intervention for adults with acquired brain injury: A pilot investigation. Neuropsychol Rehabil. 2021 Aug;31(7):1069-1090. doi: 10.1080/09602011.2020.1760892. Epub 2020 May 14. PMID 32408795